CLINICAL TRIAL: NCT04386629
Title: Evaluation of CANKADO in Breast Cancer Patients in Germany
Brief Title: Health Economy Register
Acronym: GeRA
Status: Completed | Type: Observational
Sponsor: Cankado GmbH (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20180349
Record Dates: First submitted 2020-05-04; First posted 2020-05-13 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
In breast oncology, the increasing number of oral and intravenous drug therapies pose great challenges for patient management. Numerous studies demonstrate that well-informed patients develop higher confidence in their treatment and a greater sense of disease control, resulting in increased adherence and persistence as well as potentially better outcome. The electronic Patient Reported Outcome (ePRO) tool CANKADO is designed to help oncologists to fill the gap between good, personalized care and a time and resource-saving treatment for cancer patients. CANKADO helps patients and their physicians regarding therapy management by a standardized documentation procedure and, if needed, direct feedback to patients by the integrated Pro-React system. GeRA includes patients undergoing systemic therapy for breast cancer with access to CANKADO. The trial is based on questionnaires that are answered by patients via the CANKADO Patient App. Primary objective is to gain knowledge on the health economic impact of CANKADO resource utilization in breast cancer care including the evaluation of physicians' time and patient experience.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with breast cancer
* Ongoing medical drug treatment
* 18 years or older
* CANKADO account

Exclusion Criteria:

* Lack of consent to study participation or lack of patient's ability to stuconsent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients under medical treatment for breast cancer with access to CANKADO will be included in the analysis. This study will take place in at least 10 German centers with CANKADO access / participation representatively distributed in Germany.
Sampling Method: Non-Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Occasion of consultation | 3 months
  To obtain the information on the health economic impact of CANKADO resource utilization patients will be asked to fill in a questionnaire containing a question about the occasion of consultation.
Frequency of consultation | 3 months
  To obtain the information on the health economic impact of CANKADO resource utilization patients will be asked to fill in a questionnaire containing a question about the frequency of consultation.
Duration of consultation | 3 months
  To obtain the information on the health economic impact of CANKADO resource utilization patients will be asked to fill in a questionnaire containing a question about the duration of consultation. Also, the time spent for travelling and for the appointment is included here.

SECONDARY OUTCOMES:
Quality of life (QoL): Quality of Life Questionnaire (FACT-B) | 3 months
  Quality of life (QoL) was assessed as part of the Quality of Life Questionnaire (FACT-B) as the subjective feeling of the patient
Estimate usage satisfaction of healthcare professionals: minutes | 3 months
  The usage satisfaction of healthcare professionals was evaluated by assessing the impact on workload of CANKADO assessed in minutes.
Age | 3 months
  Assessed in years
Gender | 3 months
  Assessed as male/female
Grade of education | 3 months
  Assessed as following options: secondary modern school, secondary school, abitur, university degree, promotion
Number of inhabitants in hometown | 3 months
German home state | 3 months
  Assessed as: Baden-Württemberg, Bayern, Berlin, Brandenburg, Bremen, Hamburg, Hessen, Mecklenburg-Vorpommern, Niedersachsen, Nordrhein-Westfalen, Rheinland-Pfalz, Saarland, Sachsen, Sachsen-Anhalt, Schleswig-Holstein, Thüringen
Location of treatment | 3 months
  Assessed as: university hospital, hospital, haemato-oncologist, gynaecologic oncologist
Year of primary brest cancer diagnosis | 3 months
Radiotherapy treatment of patient | 3 months
  assessed as: yes/no
Oral cancer treatment of patient | 3 months
  assessed as: yes/no
Treatment of patient with osteopretectics | 3 months
  assessed as: yes/no
Treatment of patient against high blood pressure | 3 months
  assessed as: yes/no
Treatment of patient against diabetes | 3 months
  assessed as: yes/no
Treatment of patient against asthma | 3 months
  assessed as: yes/no
employment status of patient | 3 months
  assessed as : employed, not employed, retirement

CONTACTS AND LOCATIONS:
Overall Officials: Timo Schinköthe, PhD, Study Director — Cankado GmbH
Locations (10):
- Germany (10):
  - Hämato-onkologischer Studienkreis am Klinikum Aschaffenburg, Aschaffenburg
  - Kliniken der Stadt Köln - Krankenhaus Holweide, Brustzentrum, Cologne
  - Kliniken Essen Mitte, Essen
  - Onkology Bethanien Frankfurt, Frankfurt
  - Mammazentrum Hamburg Am Krankenhaus Jerusalem, Hamburg
  - University Hospital, Mainz
  - University Hospital, Mannheim
  - University Hospital, München
  - Johanna Etienne Krankenhaus, Neuss
  - Praxisnetzwerk Hämatologie/ intern. Onkologie, Troisdorf